CLINICAL TRIAL: NCT05729893
Title: Evaluation of Post Operative Pain After Using Two Different Types of Sealers (a Randomized Clinical Trial )
Brief Title: Evaluation of Post Operative Pain After Using Two Different Types of Sealers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Sara Alsayed Endo, principal investigator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BritishUE sara
Record Dates: First submitted 2023-01-05; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients were randomly divided into two groups according to material used for obturation . each patients name will be replaced with a case number within the group to protect the privacy of medical information and data of the patients care provider and the investigator will not know the name of the patient and the assessor doesn't know the group he is assessing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resin group (Active Comparator): obturated with resin sealer
  Interventions: Other: root canal sealers
- bio ceramic group (Active Comparator): obturated with bioceramic sealer
  Interventions: Other: root canal sealers

INTERVENTIONS:
Other: root canal sealers — different sealer used in obturating root canals (resin and bio ceramic)
  Other Names: bioceramic sealer

SUMMARY:
conventional endodontic treatment is done using two different types of sealers in the obturation to evaluate the post operative pain between the two sealers

DETAILED DESCRIPTION:
STUDY WILL BE PERFORMED ON PATIENTS DIAGNOSED WITH SYMPTOMATIC IRREVERSABE PULPITIS.

TREATMENT PROTOCOL FOR ALL PATIENTS IS CONVENTIONAL ROOT CANAL TREATMENT

ACCESS CAVITY AND CLEANING AND SHAPING PROCEDURES WILL BE EXECUTED FOR ALL PATIENTS WITH THE SAME PROTOCOL

SELECTED PATIENTS WILL THEN BE DIVIDED INTO TWO GROUPS,

GROUP1: ALL CANALS WILL BE OBTURATED USING RESIN STANDARD SEALERS.

GROUP2: ALL CANALS WILL BE OBTURATED USING HIGH FLOW BIOCERAMIC SEALERS THAT ACCEPT WARM VERTICAL COMPACTION

POST OPERATIVE PAIN IN THE TWO GROUPS WILL BE EVALUATED USING THE VISUAL ANALOUG SCALE AND COMPARED AT DIFFERENT TIME PERIODS (12H, 24H, 48H, 72H)

ELIGIBILITY:
Inclusion Criteria:

* • Patients age ranges from 18-50 years old.

  * Patients with teeth diagnosed with symptomatic irreversible pulpitis.
  * Normal periapical condition confirmed by normal periapical radiograph or that with minimal widening of the PDL space
  * The teeth are restorable
  * Teeth are periodontally free.

Exclusion Criteria:

* • Teeth with immature roots

  * Non restorable teeth
  * Medically compromised patients with systemic complication that would alter the treatment.
  * Necrotic teeth
  * Teeth with apical periodontitis or periapical lesions
  * Teeth that need multiple visits treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain level comparison after root canal obturation with two different endodontic sealers: VAS (Visual Analogue Scale) at 12 hours | 12 hours
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with two different endodontic sealers: VAS (Visual Analogue Scale) at 24 hours | 24 hours
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with two different endodontic sealers: VAS (Visual Analogue Scale) at 48 hours | 48 hours
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with two different endodontic sealers: VAS (Visual Analogue Scale) at 72 hours | 72 hours
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.

CONTACTS AND LOCATIONS:
Locations (1):
- British university in egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
evaluated postoperative pain results when using different sealer types in obturation

DOCUMENTS (2):
  • Study Protocol (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT05729893/Prot_000.pdf
  • Informed Consent Form (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT05729893/ICF_001.pdf